CLINICAL TRIAL: NCT02355210
Title: Application of a Novel Synbiotic to Modulate the Human Gut Microbiota and Improve Health
Brief Title: Use of a Novel Synbiotic to Change Human Gut Bacteria and Improve Health in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Nebraska Lincoln (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USDA-NIFA-AFRI-003397
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Intestinal Microbiota and Barrier Function
MeSH Terms: interventions — 4'-galactooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): 5 g lactose given as a placebo
  Interventions: Dietary Supplement: Placebo
- Probiotic 1 (Experimental): Bifidobacteria adolescentis BD1, 10^9
  Interventions: Dietary Supplement: Bifidobacteria adolescentis BD1
- Probiotic 2 (Experimental): Bifidobacteria animalis subsp. lactis BB-12, 10^9
  Interventions: Dietary Supplement: Bifidobacteria animalis subsp. lactis BB-12
- Prebiotic (Experimental): galactooligosaccaride, 5 g
  Interventions: Dietary Supplement: galactooligosaccharide
- Synbiotic 1 (Experimental): galacto-oligosaccharide (5 g) and Bifidobacteria adolescentis BD1 (10^9)
  Interventions: Dietary Supplement: Bifidobacteria adolescentis BD1 and galactooligosaccharide
- Synbiotic 2 (Experimental): galacto-oligosaccharide (5 g) and Bifidobacteria animalis subsp. lactis BB-12 (10^9)
  Interventions: Dietary Supplement: Bifidobacteria animalis subsp. lactis BB-12 and galactooligosaccharide

INTERVENTIONS:
Dietary Supplement: Bifidobacteria adolescentis BD1 — packet containing 10^9 cells of Bifidobacteria adolescentis BD1
  Arms: Probiotic 1
Dietary Supplement: Bifidobacteria animalis subsp. lactis BB-12 — packet containing 10^9 cells of Bifidobacteria animalis subsp. lactis BB-12
  Arms: Probiotic 2
Dietary Supplement: Bifidobacteria adolescentis BD1 and galactooligosaccharide — packet containing 10^9 cells Bifidobacteria adolescentis BD1 and 5 g galactooligosaccharide
  Arms: Synbiotic 1
Dietary Supplement: Bifidobacteria animalis subsp. lactis BB-12 and galactooligosaccharide — packet containing 10^9 cells B animalis subsp. lactis BB-12 and 5 g galactooligosaccharide
  Arms: Synbiotic 2
Dietary Supplement: galactooligosaccharide — 5 g galactooligosaccharide
  Arms: Prebiotic
Dietary Supplement: Placebo — lactose powder, 5 grams
  Arms: Placebo

SUMMARY:
This study evaluates the effect of a dietary supplement to improve gut health. The participants will take one of six dietary treatments for three weeks, and the gut bacteria and the gut intestinal barrier will be assessed to determine if these dietary treatments beneficially change these markers of gut health.

DETAILED DESCRIPTION:
In this study, we intend to test the ecological and therapeutic functionality of a synbiotic combination of a Bifidobacterium adolescentis strain and the prebiotic galactooligosaccharide (GOS) in a human clinical trial. The synbiotic combination was selected based on a novel in vivo selection; specifically, the strain (BD1) is an human autochthonous gut organism that was enriched in an individual by GOS. Our experiments will test the efficacy of this synbiotic compared to a conventional synbiotic. We hypothesize this rationally selected synbiotic will improve intestinal barrier function in obese adult subjects, thereby preventing endotoxemia and metabolic inflammation, physiologically relevant functions that are increased in obese individuals. Our objectives are to: (1) compare the ability of the test and control synbiotic preparations to alter the gut microbiota in obese individuals; (2) test if GOS supports colonization and metabolic activity of test and control strains in the human gut; (3) compare the ability of the two synbiotic preparations to improve intestinal permeability and endotoxemia in obese subjects; and (4) assess associations between the gut microbiota and the test strain with biomarkers for translocation and endotoxemia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yrs, obese (30 kg/m2 and greater)

Exclusion Criteria:

* (1) prior intestinal resection, (2) patient history of GI diseases except for hiatal hernia, GERD, hemorrhoids, (3) severe renal disease defined by creatinine more than twice normal, (4) markedly abnormal liver function defined by ALT/AST over 4 times normal levels or elevated bilirubin (5) antibiotic use within the last 12 weeks prior to enrollment, (6) lean or overweight (BMI < 30 kg/m2), (7) intolerant to aspirin, (8) regular use of aspirin, (9) excessive alcohol intake (>2 drinks for men, 1 drink for women daily), (10) presence of uncontrolled chronic metabolic disease (cardiovascular disease, insulin requiring diabetes or uncontrolled diabetes, cancer, etc, (11) a plan to have a major change in dietary habit during the following 6 months, (12) consumption of probiotics, prebiotics or synbiotics without an appropriate 4 week washout period, (13) lactose intolerance or malabsorption; (14) subjects younger than 18 or older than 65, (15) unwillingness to consent to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hutkins, PhD, Principal Investigator — University of Nebraska Lincoln; Jens Walter, PhD, Principal Investigator — University of Alberta
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Krumbeck JA, Rasmussen HE, Hutkins RW, Clarke J, Shawron K, Keshavarzian A, Walter J. Probiotic Bifidobacterium strains and galactooligosaccharides improve intestinal barrier function in obese adults but show no synergism when used together as synbiotics. Microbiome. 2018 Jun 28;6(1):121. doi: 10.1186/s40168-018-0494-4. PMID 29954454

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 151 subjects enrolled. Of these, 37 subjects discontinued trial prior to treatment randomization due to loss to follow-up (n=12), subject no longer interested (n=9), laboratory values outside range (n=5), and other (n=11).
Groups:
- Prebiotic: galactooligosaccharide, 5 g
Period: Overall Study
Arm/Group | Placebo | Probiotic 1 | Probiotic 2 | Synbiotic 1 | Synbiotic 2 | Prebiotic
Started | 19 | 18 | 16 | 17 | 19 | 18
Completed | 19 | 18 | 16 | 17 | 19 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of per-protocol data presented. Thus, participant number is less than the number that completed each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Probiotic 1 | Probiotic 2 | Synbiotic 1 | Synbiotic 2 | Prebiotic | Total
Number analyzed (Participants) | 17 | 14 | 14 | 16 | 17 | 16 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (8.8) | 44.7 (13.3) | 43.9 (12.5) | 44.2 (11.8) | 43.1 (12.7) | 45.9 (9.6) | 44.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 12 | 11 | 12 | 12 | 69
  Male | 4 | 5 | 2 | 5 | 5 | 4 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 2 | 2 | 1 | 9
  Not Hispanic or Latino | 17 | 12 | 12 | 14 | 15 | 15 | 85
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 5 | 8 | 4 | 3 | 6 | 5 | 31
  Ethnicity: African American | 10 | 6 | 7 | 13 | 11 | 11 | 58
  Ethnicity: Other | 2 | 0 | 3 | 0 | 0 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 17 | 14 | 14 | 16 | 17 | 16 | 94
Education [Count of Participants; unit: Participants]
  Less than or equal to 12 years | 3 | 1 | 2 | 6 | 2 | 6 | 20
  Greater than 12 years | 14 | 13 | 12 | 10 | 15 | 10 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change in Microbiota, as Measured by Change in Microbiota Composition, Including Presence of B. Adolescentis BD1 and B. Animalis Supsp Lactis BB-12
Description: change in microbiota composition, including presence of B. adolescentis BD1 and B. animalis supsp lactis BB-12
Time Frame: baseline and three weeks
Population: Mann-Whitney-Wilcoxon matched pair tests
Measure: Mean (Standard Deviation); unit: percentage of bacterial taxa
Arm/Group | Placebo | Probiotic 1 | Probiotic 2 | Synbiotic 1 | Synbiotic 2 | Prebiotic
Number analyzed (Participants) | 17 | 14 | 14 | 16 | 17 | 16
percentage of bacterial taxa
  Bifidobacterium Baseline | 7.9 (8.1) | 9.1 (5.3) | 8.8 (5.7) | 6.0 (5.9) | 8.7 (6.2) | 11.3 (10.5)
  Bifidobacterium Treatment End | 12.0 (8.0) | 14.6 (6.9) | 9.5 (8.4) | 14.7 (7.4) | 15.9 (8.0) | 17.4 (11.4)
  OTU_1 (B adolescentis) Baseline | 1.2 (1.9) | 1.2 (4.2) | 1.2 (2.5) | 2.5 (4.5) | 3.1 (4.5) | 3.8 (7.5)
  OTU_1 (B adolescentis) Treatment End | 2.6 (4.1) | 3.4 (5.1) | 1.1 (1.6) | 7.3 (7.0) | 6.8 (9.6) | 6.6 (8.8)
  OTU_167 (B. animalis subsp. lactis) Baseline | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  OTU_167 (B. animalis subsp. lactis) Treatment End | 0.0 (0.1) | 0.0 (0.0) | 0.1 (0.1) | 0.0 (0.0) | 0.1 (0.2) | 0.2 (0.9)

2. Primary Outcome: Change in Intestinal Permeability as Measured by Change in Percent Sugars in Urine
Description: Change in intestinal permeability as measured by change in percent sugars in urine
Time Frame: baseline and three weeks
Measure: Mean (Standard Deviation); unit: sucralose:lactulose ratio
Arm/Group | Placebo | Probiotic 1 | Probiotic 2 | Synbiotic 1 | Synbiotic 2 | Prebiotic
Number analyzed (Participants) | 17 | 14 | 14 | 16 | 17 | 16
sucralose:lactulose ratio
  Sucralose:Lactulose with aspirin Baseline | 0.32 (0.20) | 0.34 (0.21) | 0.34 (0.30) | 0.32 (0.23) | 0.36 (0.19) | 0.37 (0.19)
  Sucralose:Lactulose with aspirin Treatment End | 0.36 (0.25) | 0.20 (0.16) | 0.26 (0.18) | 0.20 (0.16) | 0.29 (0.16) | 0.23 (0.15)

3. Secondary Outcome: Endotoxemia, as Measured by Change in Circulating Endotoxin by Lipopolysaccharide and Lipopolysaccharide-binding Protein
Description: Endotoxemia, as measured by change in circulating endotoxin by lipopolysaccharide and lipopolysaccharide-binding protein
Time Frame: baseline and three weeks
Measure: Mean (Standard Deviation); unit: EU/mL
Arm/Group | Placebo | Probiotic 1 | Probiotic 2 | Synbiotic 1 | Synbiotic 2 | Prebiotic
Number analyzed (Participants) | 16 | 14 | 14 | 14 | 17 | 15
EU/mL
  Lipopolysaccharide Baseline | 0.02 (0.02) | 0.03 (0.03) | 0.3 (0.03) | 0.02 (0.03) | 0.02 (0.02) | 0.02 (0.02)
  Lipopolysaccharide Treatment End | 0.02 (0.04) | 0.03 (.03) | 0.03 (0.06) | 0.02 (0.04) | 0.02 (0.02) | 0.02 (0.01)

ADVERSE EVENTS:
Arm/Group | Placebo | Probiotic 1 | Probiotic 2 | Synbiotic 1 | Synbiotic 2 | Prebiotic
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14 | 0/14 | 0/16 | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/14 | 0/16 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/14 | 0/16 | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No